CLINICAL TRIAL: NCT04862208
Title: Comparison of Fasted vs. Carbohydrate and Protein Breakfast on Exercise Metabolism and Rest of the Day Energy Intake
Brief Title: Breakfast Consumption and Energy Balance in Active Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Exercise Physiology, Ohio University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20-F-9
Record Dates: First submitted 2021-04-13; First posted 2021-04-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Energy Intake; Substrate Utilization; Hormones; Satiety
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Carbohydrate-based breakfast + exercise (Experimental): maltodextrin
  Interventions: Dietary Supplement: Maltodextrin supplement
- Protein-based breakfast + exercise (Experimental): whey
  Interventions: Dietary Supplement: Whey supplement
- Fasted breakfast + exercise (Experimental): water
  Interventions: Dietary Supplement: Water
- Carbohydrate-based breakfast + no exercise (Sham Comparator): maltodextrin
  Interventions: Dietary Supplement: Maltodextrin supplement

INTERVENTIONS:
Dietary Supplement: Maltodextrin supplement — maltodextrin (25g in 12 oz water) 1 hour pre-exercise
  Arms: Carbohydrate-based breakfast + exercise
Dietary Supplement: Whey supplement — whey (25g in 12 oz water) 1 hour pre-exercise
  Arms: Protein-based breakfast + exercise
Dietary Supplement: Water — non-caloric control (12 oz flavored water) 1 hour pre-exercise
  Arms: Fasted breakfast + exercise
Dietary Supplement: Maltodextrin supplement — maltodextrin (25g in 12 oz water) with no exercise
  Arms: Carbohydrate-based breakfast + no exercise

SUMMARY:
Exercising in the fasted state results in greater fat oxidation during exercise and results in decreased caloric intake in the meals after exercise. However, the studies that examine fasted vs. fed exercise utilize a carbohydrate-based breakfast, which can increase blood glucose and insulin concentrations, which is considered a negative consequence. A protein breakfast, which can increase satiety and rest of day energy intake could also increase resting energy expenditure as well as fat oxidation during exercise. However, comparisons between fasting exercise and pre-exercise breakfast macronutrient intake (i.e., carbohydrate vs. protein) have not been made. Therefore the purpose of this study is to investigate if eating breakfast and the composition of this breakfast before exercise has an effect on the food eaten throughout the rest of the day.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* regularly participate in exercise for at least 150 min per week
* run at least 3 days per week for 30 minutes
* able to complete a VO2max test
* able to exercise for 45 min moderate intensity exercise at one time without breaks

Exclusion Criteria:

* not participating in structured exercise of 150 min/week for the past 6 months
* not running at least 3 days per week for 30 minutes
* not attaining a VO2max of 50 ml/kg/min (60th percentile fitness classification according to the American College of Sports Medicine)
* currently smoke or quit smoking less than one year ago.
* diagnosed with or are being treated for a cardiovascular disease, high blood pressure, fibromyalgia, irritable bowel syndrome or a metabolic disorder such as diabetes, thyroid disorder, or high cholesterol.
* food allergies or sensitivities.
* not willing to have blood drawn on 4 occasions during each trial (16 total times)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in energy expenditure | immediately pre-breakfast, immediately post-breakfast, immediately pre-exercise, and immediately post-exercise
  Measured via indirect calorimetry
Change in lunch energy intake | 60 min post-exercise
  measured via standardized lunch buffet
Change in dinner energy intake | Day 1 (trial 1); between Days 6 and 8 (trial 2); between Days 11 and 15 (trial 3); and between Days 16 and 22 (trial 4)
  weight of food returned the following day
Change in appetite | immediately pre-breakfast, immediately post-breakfast, immediately post-exercise, and immediately pre-lunch
  measured via circulating hormones
Change in blood glucose | immediately pre-breakfast, immediately post-breakfast, immediately post-exercise, immediately pre-lunch, and immediately pre-dinner
  measured via fingerstick blood assessment
Change in subjective hunger | baseline, immediately pre-breakfast, immediately post-breakfast, immediately post-exercise, immediately pre-lunch, immediately post-lunch, immediately pre-dinner, and immediately post-dinner
  measured via 100mm visual analogue scale, higher scores indicate greater hunger

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No